CLINICAL TRIAL: NCT03371875
Title: Automated Youth-To-Adult Transition Planning Using Health Information ...
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, William E. Bennett, Jr., Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1704015932
Record Dates: First submitted 2017-11-17; First posted 2017-12-13 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Transition; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Clinics (Experimental): Clinics in this arm will assess the adolescent's readiness for youth-to-adult transition using the TRAQ questionnaire. Physicians will then be given reminders based on the subject's deficiencies in transition management, and given the opportunity to intervene.
  Interventions: Behavioral: Automated transition care reminders
- Control Clinics (No Intervention): Clinics in this arm will assess the adolescent's readiness for youth-to-adult transition using the TRAQ questionnaire. No reminders will be provided to providers for care transition.

INTERVENTIONS:
Behavioral: Automated transition care reminders — The CHICA system will gather the elements of the TRAQ questionnaire and report the specific areas of deficiency to the physician. If a patient reaches the point of care transition (18 years), then an automated email is sent to a clinic nurse.
  Arms: Transition Clinics

SUMMARY:
This study seeks to automate the process of youth to adult transition using an existing computerized decision support system in primary care. Subjects will complete the TRAQ readiness questionnaire after the age of 14, and then their responses will be flagged for the physician to review and provide additional transition related educational materials. Once transition is necessary, the system sends an automated email to the responsible party in the office.

DETAILED DESCRIPTION:
This proposal seeks to improve transition care using health information technology. The process of transition from a pediatric to adult provider is a universal need across both primary care and subspecialties. Little work has been done specifically within pediatric gastroenterology to address the needs of patients with chronic gastrointestinal disease. The investigators propose to use an existing computerized clinical decision support system (CHICA - the Child Health Improvement through Computer Automation system) to pilot a youth-to-adult Transition module within a large primary care network. This will be accomplished by automating the "Six Core Elements of Healthcare Transition" set forth by the National Health Care Transition Center. These core elements consist of: (1) sharing the transition policy with families, (2) providing transition tracking and monitoring, (3) assessing transition readiness using a standardized tool (the TRAQ - Transition Readiness Assessment Questionnaire), (4) transition planning through iterative preparation of all necessary transition skills and documents, (5) accomplishing the transfer of care itself, and (6) assessing transfer completion. Each of these core elements will be accomplished using a combination of patient-facing (tablets) and providerfacing (webforms alongside the electronic medical record). Once these software rules are written and tested, they will be piloted in the existing primary care decision support system. The investigators will iteratively assess the following goals: (1) each patient's transition readiness as appropriate for their age, and (2) provider and patient satisfaction with the transition process. These outcomes will be compared in a prepost design, data will be collected during the first 6 months prior to the Transition module being implemented in CHICA. Following this 6-month period, the Transition module will be turned on, and a repeat assessment made of these outcomes. If this pilot test is successful, the investigators will then be ready to launch this module in a similar system (CHICA-GI) that will be live in the pediatric gastroenterology clinic. Once this system has a transition module active, the investigators will be able to test if it accomplishes similar goals for gastroenterology subspecialty patients, including disease-specific transition goals, in future R21 and R01 applications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 14-18 (those who need transition) and seen at an Eskenaki pediatrics clinic in past month.

Exclusion Criteria:

* None.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Patient transition satisfaction (Pre) | Baseline
  Families will be called by study RA and asked the following questions:
  Has your pediatrician shared with you (your child) their clinic's approach to transitioning you from pediatric to adult health care? Have you (or your child) ever been asked to complete a survey at your pediatrician's office regarding your health and how to use health care? Did you and your pediatric provider talk about you being more in charge of your health? Did you and this provider talk about you scheduling your own appointments with this provider instead of your parent or guardian? Did you and this provider talk about how your health insurance might change as you get older? Did you and this provider talk about whether you may need to change to a new provider who treats mostly adults? Did this provider ask if you had any questions or concerns about changing to a new provider who treats mostly adults?
Patient transition satisfaction (Post) | 1 month after appointment
  Families will be called by study RA and asked the following questions:
  Has your pediatrician shared with you (your child) their clinic's approach to transitioning you from pediatric to adult health care? Have you (or your child) ever been asked to complete a survey at your pediatrician's office regarding your health and how to use health care? Did you and your pediatric provider talk about you being more in charge of your health? Did you and this provider talk about you scheduling your own appointments with this provider instead of your parent or guardian? Did you and this provider talk about how your health insurance might change as you get older? Did you and this provider talk about whether you may need to change to a new provider who treats mostly adults? Did this provider ask if you had any questions or concerns about changing to a new provider who treats mostly adults?

SECONDARY OUTCOMES:
Provider satisfaction | 6 months
  A Likert scale is administered twice yearly determining the provider satisfaction with each CHICA module

CONTACTS AND LOCATIONS:
Overall Officials: William E Bennett, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided